CLINICAL TRIAL: NCT04932499
Title: Can Mindfulness Meditation Reduce Peri-Operative Pain and Anxiety Following Total Joint Arthroplasty?
Brief Title: Mindfulness Meditation for Surgical Pain and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Farrah Morrow, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mindfulness Study
Record Dates: First submitted 2021-06-04; First posted 2021-06-21 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
Keywords: Total Hip Arthroplasty; Mindfulness Meditation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Standard of Care; Mindfulness

STUDY DESIGN:
Intervention Model Description: Single blinded, block randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard of care
  Interventions: Other: Standard of Care
- Mindfulness Meditation (Experimental): Mindfulness meditation in addition to standard of care
  Interventions: Other: Standard of Care; Other: Mindfulness Meditation

INTERVENTIONS:
Other: Standard of Care — Participants randomly assigned to this intervention will receive standard of care given to all patients undergoing total knee arthroplasty at our institution as outlined in the Common Care Pathway for Total Joint Replacement. Outcome assessments will be completed pre-operatively, each day while in hospital and 7 and 14 days postoperative.
Other: Mindfulness Meditation — In addition to standard of care, participants randomly assigned to the treatment group will be given a 45-60 minute teaching session on mindfulness meditation. Upon completion of this session, participants will be given "homework" recordings of a body scan exercise and asked to listen to the recording daily for the two-week period prior to surgery. Participants will be asked to listen to their recording immediately prior to their surgery and daily while in hospital. In addition, participants assigned to mindfulness intervention will receive standard of care as outlined in the control group. Outcome assessments will be completed pre-operatively, each day while in hospital and 7 and 14 days postoperative.
  Arms: Mindfulness Meditation

SUMMARY:
Health care professionals are dedicated to the ongoing evaluation of the peri-operative experience, and always striving to improve patient satisfaction. There are extensive protocols and communication strategies to optimize pre-operative education, intra-operative comfort and safety, and post-operative pain control, but most strategies are carried out by the treating team. The idea of using mindfulness to empower patients to be active participants in reducing pain and anxiety has already been successful in a number of medical settings.

Multiple studies have demonstrated the effectiveness of mindfulness based stress reduction and mindfulness based cognitive therapy, a modification to treat depression. Mindfulness has been shown to reduce catastrophizing, depression and disability, all of which are of concern with respect to long-term success after arthroplasty. There is limited evidence to demonstrate the usefulness of mindfulness as a peri-operative intervention. Although there is evidence that a brief mindfulness meditation session can impact experimental pain scores and anxiety, there is no current literature that has evaluated the impact of such a session as part of the peri-operative teaching protocol with respect to pain and anxiety.

Our objective is to assess the capability of a short-term mindfulness intervention (serving as a compliment to the pre-operative pathway for total joint arthroplasty) to reduce peri-operative pain that can be integrated with the existing arthroplasty pathway. In addition, we explore the utility of using such a tool to reframe patients' expectation of the peri-operative period as evidence by its impact on anxiety and post-operative patient satisfaction.

Thirty-two participants will be recruited and randomly assigned to either control or treatment groups. The control group will receive standard care associated with total joint arthroplasty. The treatment group will receive a 45-60 minute mindfulness meditation teaching session administered by a credentialed mindfulness instructor and affiliated with the University of Calgary Psychosocial Oncology Mindfulness Program in addition to standard care for arthroplasty surgery. The treatment group will be assigned "homework" recordings of body scan exercises and asked to listen to the recording daily for the two-week period prior to surgery. Patients will be asked to listen to their body scan meditation immediately prior to entering the operating room and daily each post-operative day while in hospital. Longitudinal assessments encompassing the preoperative, peri-operative and post-operative periods will be acquired using validated pain scores and anxiety outcomes scores including the Numerical Rating Scale (NRS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the short-form State-Trait Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* elective total knee arthroplasty

Exclusion Criteria:

* non-English speaking
* patients requiring general anesthesia
* psychiatric illness
* chronic pain requiring > 8 tablets per day of tramacet, Tylenol #3 or Percocet
* joint revision surgery
* patients who meet criteria for acute pain service stratification and referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale (NRS) pain scores | day of surgery; daily as inpatient; 7 days postoperative; 14 days postoperative
  Longitudinal assessment of Numerical Rating Scale (NRS) pain scores. Scale ranges from 0-10 with 0 representative of no pain to 10 worst pain possible

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | day of surgery; daily as inpatient; 7 days postoperative; 14 days postoperative
  Longitudinal assessment of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Individual test questions are scored on a scale from 0-4 with 0 representing "none" to 4 representing "extreme". Total score is 96 with a higher score representing more pain, increased stiff, decreased physical function
Change in Anxiety Scores | day of surgery; daily as inpatient; 7 days postoperative; 14 days postoperative
  Longitudinal assessment of short-form State-Trait Anxiety Inventory (STAI). This assessment consists of six questions with scores ranging from 6 to 24 (high score representative of increased anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- South Health Campus, Calgary, Alberta, Canada